CLINICAL TRIAL: NCT04627467
Title: Prophylaxis With Chloroquine in Health Personnel Exposed to Infection With Coronavirus Disease 2019 (COVID-19)
Brief Title: Prevention With Chloroquine in Health Personnel Exposed to Infection With Coronavirus Disease 2019 (COVID-19) (TS-COVID)
Acronym: TS-COVID
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundacion Clinica Valle del Lili (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: FVL-1567
Record Dates: First submitted 2020-10-30; First posted 2020-11-13 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2020-09

CONDITIONS: Covid19
Keywords: Chloroquine; COVID-19; SARS-CoV-2; Antibodies; Prophylaxis; Healthcare workers
MeSH Terms: conditions — COVID-19 | interventions — Chloroquine

STUDY DESIGN:
Intervention Model Description: Single arm study in which healthcare workers were actively invited to participate. After verifying volunteer's eligibility through a survey that evaluated the presence of COVID-19 symptoms (primary efficacy outcome), 150 mg chloroquine base was dispensed in site by a pharmaceutical chemist at days 0, 15, 30, 45, 60, and 75. Questions regarding adverse drugs reactions (safety outcome) were included in the survey after the first dose was administered. Participants who discontinued chloroquine were followed up until study completion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chloroquine 150mg base (Experimental): Volunteers received chloroquine tablets orally at days 0, 15, 30, 45, 60 and 75.
  Interventions: Drug: Chloroquine

INTERVENTIONS:
Drug: Chloroquine — 250mg tablet (150mg base chloroquine)

SUMMARY:
The purpose of this study is to assess the efficacy and safety of chloroquine prophylaxis on the incidence of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) infections in healthcare workers exposed to patients with confirmed Coronavirus Disease 2019 (COVID-19)

DETAILED DESCRIPTION:
Single arm study in which healthcare workers were actively invited to participate. Possible participants were asked to complete a questionnaire to determine eligibility for study entry and to identify risk factors for infection, severe infection, or adverse events associated with chloroquine use.

Volunteers who meet the eligibility requirements received chloroquine 150mg base at days 0, 15, 30, 45, 60, 75. Cumulative incidence and incidence rate of COVID-19 at days 30,60 and 90 were calculated. Presence of Immunoglobulin G (IgG) antibodies against SARS-Cov-2 was evaluated at the beginning, at the end and at any moment if they become infected with this virus.

In addition, patients were asked to complete a survey evaluating adverse effects and COVID-19 symptoms at day 0 and weeks 2,4,6,8,10, and 12.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic healthcare workers and contractors who work in Fundacion Valle del Lili

Exclusion Criteria:

* To have two or more of the following symptoms 14 days previous to the initial assessment: cough, dyspnea, odynophagia, fatigue, weakness, fever >38 degrees °C
* History of close contact (less than two meters) with a person with probable or confirmed COVID-19 without adequate protection during the last 14 days
* History of one the following diseases in treatment at inclusion in the study: cardiac arrhythmias, epilepsy, kidney disease, seizures
* Treatment with concomitant medications: tamoxifen, quinine, cyclosporine, amiodarone, digoxine, anticonvulsivants
* Having recently taken chloroquine or hydroxychloroquine in the last two weeks
* Known hypersensitivity to chloroquine or hydroxychloroquine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3217 (Actual)
Dates: Start 2020-03-28 (Actual); Primary Completion 2020-07-09 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
COVID-19 infection | Day 15
  Symptomatic COVID-19 infection confirmed by reverse transcriptase polymerase chain reaction in healthcare workers, in any respiratory sample
COVID-19 infection | Day 30
  Symptomatic COVID-19 infection confirmed by reverse transcriptase polymerase chain reaction in healthcare workers, in any respiratory sample
COVID-19 infection | Day 45
  Symptomatic COVID-19 infection confirmed by reverse transcriptase polymerase chain reaction in healthcare workers, in any respiratory sample
COVID-19 infection | Day 60
  Symptomatic COVID-19 infection confirmed by reverse transcriptase polymerase chain reaction in healthcare workers, in any respiratory sample
COVID-19 infection | Day 75
  Symptomatic COVID-19 infection confirmed by reverse transcriptase polymerase chain reaction in healthcare workers, in any respiratory sample
COVID-19 infection | Day 90
  Symptomatic COVID-19 infection confirmed by reverse transcriptase polymerase chain reaction in healthcare workers, in any respiratory sample

SECONDARY OUTCOMES:
IgG antibodies seropositivity against SARS-CoV-2 | Day 90
  Number of participants with IgG antibodies seropositivity against SARS-CoV-2 in the final sample.

OTHER OUTCOMES:
Adverse drug event | Day 15, day 30, day 45, day 60, day 75 and day 90
  Number of participants with at least one adverse drug event
Unexpected adverse events | Day 15, day 30, day 45, day 60, day 75 and day 90
  Number of participants with unexpected adverse events
Participant drop-out | Baseline and day 90
  Number of participants who did not completed prophylaxis because of discontinuing medication, withdrawal of consent, or lost to follow-up
Non-adherence | Baseline and day 90
  Number of participants who were not-adherent to the medication scheme

CONTACTS AND LOCATIONS:
Overall Officials: Juan D Velez, MD, Principal Investigator — Fundacion Clinica Valle del Lili
Locations (1):
- Fundacion Valle del Lili, Cali, Valle del Cauca Department, Colombia

IPD SHARING:
Plan to Share IPD: No
We do not plan to share IPD, since we are not allowed to share information concerning medical history of our patients or health workers.

REFERENCES:
- [Result] WHO. Coronavirus disease 2019 (COVID-19). Situation Report - 43 2020 [Available from: https://www.who.int/emergencies/diseases/novel-coronavirus2019/technicalguidance/laboratoryguidance
- [Result] Wang M, Su S, Lv J, Zhou G, Wang Q, Guo C. Analysis of clinical features and prognostic factors in Chinese patients with rheumatic diseases in an intensive care unit. The Egyptian Rheumatologist. 2018;40(1):63-6.
- [Result] Livingston E, Bucher K. Coronavirus Disease 2019 (COVID-19) in Italy. JAMA. 2020 Apr 14;323(14):1335. doi: 10.1001/jama.2020.4344. No abstract available. PMID 32181795
- [Result] Wang M, Cao R, Zhang L, Yang X, Liu J, Xu M, Shi Z, Hu Z, Zhong W, Xiao G. Remdesivir and chloroquine effectively inhibit the recently emerged novel coronavirus (2019-nCoV) in vitro. Cell Res. 2020 Mar;30(3):269-271. doi: 10.1038/s41422-020-0282-0. Epub 2020 Feb 4. No abstract available. PMID 32020029
- [Result] Gautret P, Lagier JC, Parola P, Hoang VT, Meddeb L, Mailhe M, Doudier B, Courjon J, Giordanengo V, Vieira VE, Tissot Dupont H, Honore S, Colson P, Chabriere E, La Scola B, Rolain JM, Brouqui P, Raoult D. RETRACTED: Hydroxychloroquine and azithromycin as a treatment of COVID-19: results of an open-label non-randomized clinical trial. Int J Antimicrob Agents. 2020 Jul;56(1):105949. doi: 10.1016/j.ijantimicag.2020.105949. Epub 2020 Mar 20. PMID 32205204
- [Result] Zhou D, Dai SM, Tong Q. COVID-19: a recommendation to examine the effect of hydroxychloroquine in preventing infection and progression. J Antimicrob Chemother. 2020 Jul 1;75(7):1667-1670. doi: 10.1093/jac/dkaa114. PMID 32196083
- [Result] Rodriguez-Morales AJ, Cardona-Ospina JA, Gutierrez-Ocampo E, Villamizar-Pena R, Holguin-Rivera Y, Escalera-Antezana JP, Alvarado-Arnez LE, Bonilla-Aldana DK, Franco-Paredes C, Henao-Martinez AF, Paniz-Mondolfi A, Lagos-Grisales GJ, Ramirez-Vallejo E, Suarez JA, Zambrano LI, Villamil-Gomez WE, Balbin-Ramon GJ, Rabaan AA, Harapan H, Dhama K, Nishiura H, Kataoka H, Ahmad T, Sah R; Latin American Network of Coronavirus Disease 2019-COVID-19 Research (LANCOVID-19). Electronic address: https://www.lancovid.org. Clinical, laboratory and imaging features of COVID-19: A systematic review and meta-analysis. Travel Med Infect Dis. 2020 Mar-Apr;34:101623. doi: 10.1016/j.tmaid.2020.101623. Epub 2020 Mar 13. PMID 32179124
- [Result] Xu X, Yu C, Qu J, Zhang L, Jiang S, Huang D, Chen B, Zhang Z, Guan W, Ling Z, Jiang R, Hu T, Ding Y, Lin L, Gan Q, Luo L, Tang X, Liu J. Imaging and clinical features of patients with 2019 novel coronavirus SARS-CoV-2. Eur J Nucl Med Mol Imaging. 2020 May;47(5):1275-1280. doi: 10.1007/s00259-020-04735-9. Epub 2020 Feb 28. PMID 32107577
- [Result] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Result] Gostic K, Gomez AC, Mummah RO, Kucharski AJ, Lloyd-Smith JO. Estimated effectiveness of symptom and risk screening to prevent the spread of COVID-19. Elife. 2020 Feb 24;9:e55570. doi: 10.7554/eLife.55570. PMID 32091395
- [Result] Chowell G, Abdirizak F, Lee S, Lee J, Jung E, Nishiura H, Viboud C. Transmission characteristics of MERS and SARS in the healthcare setting: a comparative study. BMC Med. 2015 Sep 3;13:210. doi: 10.1186/s12916-015-0450-0. PMID 26336062
- [Result] Epidemiology Working Group for NCIP Epidemic Response, Chinese Center for Disease Control and Prevention. [The epidemiological characteristics of an outbreak of 2019 novel coronavirus diseases (COVID-19) in China]. Zhonghua Liu Xing Bing Xue Za Zhi. 2020 Feb 10;41(2):145-151. doi: 10.3760/cma.j.issn.0254-6450.2020.02.003. Chinese. PMID 32064853
- [Result] Su A. Doctors and nurses fighting coronavirus in China die of both infection and fatigue. Los Angeles Times. 2020.
- [Result] Liu M, He P, Liu HG, Wang XJ, Li FJ, Chen S, Lin J, Chen P, Liu JH, Li CH. [Clinical characteristics of 30 medical workers infected with new coronavirus pneumonia]. Zhonghua Jie He He Hu Xi Za Zhi. 2020 Feb 17;43(0):E016. doi: 10.3760/cma.j.issn.1001-0939.2020.0016. Online ahead of print. Chinese. PMID 32062957
- [Result] Mitja O, Clotet B. Use of antiviral drugs to reduce COVID-19 transmission. Lancet Glob Health. 2020 May;8(5):e639-e640. doi: 10.1016/S2214-109X(20)30114-5. Epub 2020 Mar 19. No abstract available. PMID 32199468
- [Result] Welliver R, Monto AS, Carewicz O, Schatteman E, Hassman M, Hedrick J, Jackson HC, Huson L, Ward P, Oxford JS; Oseltamivir Post Exposure Prophylaxis Investigator Group. Effectiveness of oseltamivir in preventing influenza in household contacts: a randomized controlled trial. JAMA. 2001 Feb 14;285(6):748-54. doi: 10.1001/jama.285.6.748. PMID 11176912
- [Result] Hydroxychloroquine Chemoprophylaxis in Healthcare Personnel in Contact With COVID-19 Patients (PHYDRA Trial) - Full Text View. ClinicalTrials.gov.
- [Result] Chloroquine Prevention of Coronavirus Disease (COVID-19) in the Healthcare Setting - Full Text View. ClinicalTrials.gov
- [Result] Treatment of COVID-19 Cases and Chemoprophylaxis of Contacts as Prevention - Full Text View. ClinicalTrials.gov
- [Result] Ruiz-Irastorza G, Ramos-Casals M, Brito-Zeron P, Khamashta MA. Clinical efficacy and side effects of antimalarials in systemic lupus erythematosus: a systematic review. Ann Rheum Dis. 2010 Jan;69(1):20-8. doi: 10.1136/ard.2008.101766. PMID 19103632
- [Result] Kuznik A, Bencina M, Svajger U, Jeras M, Rozman B, Jerala R. Mechanism of endosomal TLR inhibition by antimalarial drugs and imidazoquinolines. J Immunol. 2011 Apr 15;186(8):4794-804. doi: 10.4049/jimmunol.1000702. Epub 2011 Mar 11. PMID 21398612
- [Result] Savarino A, Boelaert JR, Cassone A, Majori G, Cauda R. Effects of chloroquine on viral infections: an old drug against today's diseases? Lancet Infect Dis. 2003 Nov;3(11):722-7. doi: 10.1016/s1473-3099(03)00806-5. PMID 14592603
- [Result] Yan Y, Zou Z, Sun Y, Li X, Xu KF, Wei Y, Jin N, Jiang C. Anti-malaria drug chloroquine is highly effective in treating avian influenza A H5N1 virus infection in an animal model. Cell Res. 2013 Feb;23(2):300-2. doi: 10.1038/cr.2012.165. Epub 2012 Dec 4. No abstract available. PMID 23208422
- [Result] IDOATE A, IDOIPE Á. 2.4. Investigación y ensayos clínicos.
- [Result] Schwartz E. Prophylaxis of malaria. Mediterr J Hematol Infect Dis. 2012;4(1):e2012045. doi: 10.4084/MJHID.2012.45. Epub 2012 Jun 29. PMID 22811794
- [Result] Gozal D, Hengy C, Fadat G. Prolonged malaria prophylaxis with chloroquine and proguanil (chloroguanide) in a nonimmune resident population of an endemic area with a high prevalence of chloroquine resistance. Antimicrob Agents Chemother. 1991 Feb;35(2):373-6. doi: 10.1128/AAC.35.2.373. PMID 2024970
- [Result] Yao X, Ye F, Zhang M, Cui C, Huang B, Niu P, Liu X, Zhao L, Dong E, Song C, Zhan S, Lu R, Li H, Tan W, Liu D. In Vitro Antiviral Activity and Projection of Optimized Dosing Design of Hydroxychloroquine for the Treatment of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2). Clin Infect Dis. 2020 Jul 28;71(15):732-739. doi: 10.1093/cid/ciaa237. PMID 32150618
- [Result] Chen W, Huang Y. To Protect Health Care Workers Better, To Save More Lives With COVID-19. Anesth Analg. 2020 Jul;131(1):97-101. doi: 10.1213/ANE.0000000000004834. PMID 32541583